CLINICAL TRIAL: NCT07183462
Title: Azithromycin and Ampicillin for Late PPROM
Acronym: ALPRO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-1755-24-NG-CTIL; MOH_2025-04-30_014029 (Other: MOH)
Record Dates: First submitted 2025-06-04; First posted 2025-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Complications, Infectious; Premature Birth; Neonatal Diseases and Abnormalities; Antibiotic Prophylaxis; Latency Period; Prematurity
MeSH Terms: conditions — Pregnancy Complications, Infectious; Premature Birth; Congenital, Hereditary, and Neonatal Diseases and Abnormalities | interventions — Ampicillin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups. One group receives the standard antibiotic regimen, while the other group receives the standard regimen plus a single dose of intravenous Azithromycin. Both groups are followed concurrently to compare outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard antibiotic regimen (Ampicillin and Amoxicillin) (Active Comparator): Participants in the control arm receive the standard antibiotic regimen for late PPROM, consisting of intravenous Ampicillin 2g every 6 hours for 48 hours, followed by oral Amoxicillin 500mg every 8 hours for 5 days, administered according to current clinical guidelines
  Interventions: Drug: Ampicillin/Amoxicillin plus single-dose PO Azithromycin
- Intervention Arm - Standard Antibiotics with Azithromycin (Experimental): Participants in this arm will receive the standard antibiotic regimen of intravenous Ampicillin followed by oral Amoxicillin, plus a single dose of 1 gram oral Azithromycin
  Interventions: Drug: Intravenous Ampicillin followed by Oral Amoxicillin

INTERVENTIONS:
Drug: Intravenous Ampicillin followed by Oral Amoxicillin — This intervention consists of intravenous Ampicillin 2 grams every 6 hours for 48 hours, followed by oral Amoxicillin 500 mg every 8 hours for 5 days
  Arms: Intervention Arm - Standard Antibiotics with Azithromycin
Drug: Ampicillin/Amoxicillin plus single-dose PO Azithromycin — This intervention includes intravenous Ampicillin 2 grams every 6 hours for 48 hours, followed by oral Amoxicillin 500 mg every 8 hours for 5 days, plus a single dose of oral Azithromycin 1 gram administered once at the start of treatment
  Arms: Standard antibiotic regimen (Ampicillin and Amoxicillin)

SUMMARY:
The goal of this clinical trial is to learn whether adding azithromycin to the standard antibiotic treatment (ampicillin) improves newborn outcomes in women with preterm premature rupture of membranes (PPROM) between 34.0 and 36.6 weeks of pregnancy.

The main question it aims to answer is:

Does the combination of ampicillin and azithromycin lower the risk of serious neonatal health problems compared to ampicillin alone?

Researchers will compare two antibiotic regimens:

Ampicillin alone, which is the current standard care Ampicillin with azithromycin, a broader regimen that may better prevent infections and prolong pregnancy

Participants will:

Receive one of the two antibiotic treatments during hospitalization. Be monitored until delivery for signs of infection and labor

All participants will stay in the hospital until delivery. The study also looks at how the antibiotic choice may affect the time between membrane rupture and delivery, maternal infections, and the need for neonatal intensive care.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) occurs in 1-3% of all pregnancies and accounts for approximately 30% of all preterm births. It is associated with significant maternal, fetal, and neonatal risks, including infections, respiratory complications, and adverse neurodevelopmental outcomes. The management of PPROM before 34 weeks is well established and includes corticosteroids and antibiotic therapy to prolong latency and reduce infectious complications. However, optimal management of PPROM in the late preterm period (34.0 to 36.6 weeks) remains under debate.

Historically, immediate delivery was recommended after PPROM at 34 weeks or later. More recent evidence, however, suggests that expectant management may reduce neonatal respiratory morbidity, mechanical ventilation, and NICU stays, even in the late preterm period. As a result, expectant management has become more accepted. In this setting, prophylactic antibiotics are commonly used to reduce maternal and neonatal infections. While ampicillin is the standard agent used for GBS prophylaxis, it is unclear whether broader antibiotic coverage might lead to better neonatal outcomes by delaying delivery or preventing ascending infections.

In early preterm PPROM (<32 weeks), a combination of ampicillin and erythromycin (or azithromycin) has demonstrated improved outcomes in large trials. However, few studies have addressed the benefits of such regimens in late PPROM, and no randomized controlled trials to date have compared different antibiotic regimens in this specific population.

This multicenter randomized controlled trial will compare two antibiotic regimens in women with PPROM between 34.0 and 36.6 weeks of gestation:

Control group (standard care): Intravenous ampicillin 2 g every 6 hours for 48 hours, followed by oral amoxicillin 500 mg every 8 hours for 5 days.

Intervention group: Same regimen as the control group, with the addition of a single dose of PO azithromycin 1 g administered at the start of treatment.

The primary outcome is a composite of neonatal adverse outcomes, including:

Use of respiratory support (CPAP, HFNC, mechanical ventilation, ECMO) Neonatal sepsis (confirmed by positive blood culture) Hypoglycemia requiring treatment Hyperbilirubinemia requiring phototherapy Stillbirth or neonatal death within 72 hours

Secondary neonatal outcomes include:

Components of the primary outcome analyzed individually RDS, need for resuscitation, surfactant use, TTN, IVH, NEC, NICU stay duration, pneumothorax, asphyxia, convulsions, placental pathology, and others Maternal outcomes include Latency from randomization to delivery Chorioamnionitis, fever, bacteremia, placental abruption, cesarean delivery Composite maternal morbidity Postpartum infections, need for ICU admission, wound complications Length of postpartum hospital stay and breastfeeding initiation

Participants will be hospitalized from diagnosis until delivery. Management will include:

Regular maternal vital signs and infection monitoring Twice-daily fetal heart rate monitoring Corticosteroids for fetal lung maturation (in selected patients) Ultrasound to assess fetal well-being No tocolysis will be administered Labor will be induced at 37 weeks or earlier if indicated

Inclusion criteria:

Women aged 18-50 years with singleton pregnancy PPROM diagnosed between 34.0 and 36.6 weeks No active labor or signs of infection at presentation

Exclusion criteria:

Multiple gestation, chorioamnionitis, abnormal fetal heart rate, cerclage, meconium-stained amniotic fluid, fetal malformations, or GBS macrolide allergy Diagnosis of PPROM will be based on history and physical exam, including pooling seen on sterile speculum exam. When necessary, AmniSure testing will confirm membrane rupture.

Eligible women will be approached within 24 hours of admission. After obtaining informed consent, participants will be randomized (1:1) and stratified by center and gestational age (<35 weeks or ≥35 weeks). Women will remain inpatients until delivery, and labor will be induced no later than 37.0 weeks, unless earlier delivery is indicated.

Placental pathology and culture will be performed in all participants after delivery.

The sample size is based on an expected 50% rate of the composite neonatal outcome in the control group. A total of 296 women will provide 80% power to detect a 33% relative reduction in the primary outcome (from 50% to 33.5%) with a 5% alpha level. Including a 5% loss to follow-up, 311 women will be enrolled.

Data will be collected using REDCap, and participant confidentiality will be maintained through study ID numbers. Results may be used in future research but will remain de-identified.

Ethics approval will be obtained at each participating site. All participants will provide written informed consent, and the study will be conducted under standard GCP (Good Clinical Practice) guidelines.

This trial aims to provide the first direct comparison of two antibiotic regimens in the setting of late preterm PPROM, potentially impacting future recommendations on latency antibiotic therapy and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 18-50
* Premature rupture of membranes
* Gestational age 34.0 and 36.4 weeks
* Singleton pregnancy

Exclusion Criteria:

* Multiple gestations
* Individuals in active labor (defined as 3 cm dilatation and 80% effacement or more. or regular uterine construction of more than 4 in 10 minutes)
* Meconium stain amniotic fluid
* Non-reassuring fetal heart rate or status
* Maternal or fetal indication for labor:

  * Suspected Chorioamnionitis
  * Suspected placental abruption
  * Any maternal morbidity requiring labor
* Cervical cerclage in place.
* Major fetal malformation or known chromosomal abnormalities.
* Stillbirth.
* Sensitivity to Macrolides Antibiotics

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is based on biological sex (female) and pregnancy status with PPROM between 34.0 and 36.6 weeks of gestation, irrespective of the participant's gender identity
Enrollment: 311 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
A composite of neonatal adverse outcomes | From the time of birth until 72 hours postpartum
  A composite of neonatal adverse outcomes defined as the occurrence of one or more of the following events within 72 hours after birth:
  use of continuous positive airway pressure (CPAP) or high-flow nasal cannula, supplemental oxygen with a fraction of inspired oxygen (FiO2) ≥0.30 for ≥4 continuous hours, extracorporeal membrane oxygenation (ECMO), mechanical ventilation, neonatal sepsis (defined as positive blood culture), hypoglycemia requiring treatment, hyperbilirubinemia requiring phototherapy, stillbirth, or neonatal death within 72 hours after delivery
  The composite will be reported as the number of infants who experience at least one of the listed adverse outcomes.
  Unit of Measure: Number of infants with ≥1 adverse outcome

SECONDARY OUTCOMES:
Number of Infants With Severe Respiratory Morbidity | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first.
  Includes infants requiring CPAP or high-flow nasal cannula for ≥12 hours or mechanical ventilation, or neonatal death
Number of Infants Requiring Resuscitation at Birth | At birth
  Any newborn requiring active resuscitation immediately after birth
Number of Infants Diagnosed With Respiratory Distress Syndrome | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Based on clinical signs, FiO₂ >0.21, and characteristic chest X-ray findings
Number of Infants Receiving Surfactant Therapy | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first.
  Administration of surfactant during hospitalization
Number of Infants Diagnosed With Transient Tachypnea of the Newborn | Within first 72 hours after birth
  Tachypnea resolving within 72 hours after birth
Number of Infants Diagnosed With Necrotizing Enterocolitis | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first.
  Clinical diagnosis of NEC during hospitalization
Number of Infants With Grade 3 or 4 Intraventricular Hemorrhage | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first.
  Diagnosed by cranial ultrasound or imaging during hospitalization
Number of Infants With Feeding Intolerance | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first.
  Clinical diagnosis of feeding intolerance during hospitalization
Number of Infants With NICU Stay Exceeding 3 Days | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Length of NICU admission greater than three days
Number of Infants Diagnosed With Pneumothorax | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Radiologically confirmed pneumothorax during hospitalization
Number of Infants Diagnosed With Meconium Aspiration Syndrome | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Clinical diagnosis during hospitalization
Number of Infants Diagnosed With Birth Asphyxia | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Clinical diagnosis of perinatal asphyxia during hospitalization
Number of Infants Diagnosed With Periventricular Leukomalacia | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Diagnosed by imaging during hospitalization
Number of Infants With Neonatal Convulsions | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Clinically diagnosed seizures during hospitalization
Number of Neonatal Deaths | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Death of the newborn during hospitalization
Distribution of Placental Histopathology Lesion Types | Within 6 weeks after delivery, upon receipt of pathology results
  Classification of placental lesions according to standardized pathology criteria, including maternal vascular malperfusion lesions, fetal vascular malperfusion lesions, inflammatory lesions, and other abnormalities. Each placenta will be categorized based on pathology report
Number of Infants With Positive Placental Cultures | Within 6 weeks after delivery, upon receipt of culture results
  Number of infants whose placental tissue culture was positive for bacterial growth
Distribution of Bacterial Species in Positive Placental Cultures | Within 4 weeks after delivery, upon receipt of culture results
  Identification and classification of bacterial species isolated from positive placental tissue cultures. Each positive culture will be categorized by bacterial genus and speciesWithin 4 weeks after delivery, upon receipt of culture results
Latency From Randomization to Delivery | From randomization until delivery
  Number of days from randomization until delivery
Number of Participants Completing Full Course of Antenatal Corticosteroids | From randomization until delivery
  Completion of full corticosteroid course for fetal lung maturity
Number of Participants With Placental Abruption | From randomization until delivery
  Clinically diagnosed placental abruption
Number of Participants With Intrapartum Fever (≥ 38°C) | During labor
  Maternal fever occurring during labor
Number of Participants Diagnosed With Clinical Chorioamnionitis | From randomization until delivery
  Diagnosis based on uterine tenderness and/or maternal fever related to suspected uterine infection
Number of Participants With Bacteremia (Positive Blood Culture) | From randomization until 72 hours postpartum
  Positive maternal blood cultures indicating bacteremia
Number of Participants Undergoing Unplanned Cesarean Delivery | From randomization until delivery
  Cesarean delivery not planned before labor onset
Number of Participants With Postpartum Endometritis | From delivery until 6 weeks post partum
  Clinical diagnosis of postpartum endometritis
Number of Participants With Postpartum Wound Infection or Dehiscence | from birth and up to 6 weeks postpartum
  Clinical diagnosis of wound infection or dehiscence after delivery
Number of Participants With Composite Adverse Maternal Outcome | From randomization until 6 weeks postpartum
  A composite of maternal adverse outcomes defined as the occurrence of one or more of the following events within 6 weeks postpartum: bacteremia, ICU admission, hysterectomy, or need for drainage or relaparotomy
Length of Postpartum Hospital Stay | From delivery through neonatal hospitalization or up to 28 days of life, whichever comes first
  Number of days hospitalized postpartum
Number of Participants Who Initiated Breastfeeding | From delivery through maternal hospital discharge or up to 28 days postpartum, whichever comes first
  Initiation of breastfeeding during hospital stay
Number of Participants Requiring Hospital Readmission | Up to 6 weeks postpartum
  Any hospital readmission within 6 weeks postpartum
Number of Participants With Antepartum Hemorrhage | From randomization until delivery
  Clinically diagnosed bleeding before delivery
Number of Participants With Uterine Rupture | During labor or delivery
  Clinically diagnosed uterine rupture during labor or delivery
Number of Participants With Umbilical Cord Prolapse | From randomization until delivery
  Clinically diagnosed cord prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Noa Gonen, MD, Study Chair — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT07183462/Prot_000.pdf